CLINICAL TRIAL: NCT07265635
Title: Functional Proteomics of Uremic Retention Solutes Associated With Immunosenescence, Inflammation and Impaired Adaptive Stress Response
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Carmelo Libetta, Carmelo Libetta, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PROTEURS
Record Dates: First submitted 2025-11-14; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-08

CONDITIONS: Hemodialysis

STUDY DESIGN:
Intervention Model Description: This is a monocentric, randomized, controlled, crossover trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- patients on regular hemodialysis (HD) HDF with high cut-off polymethylmethacrylate (PMMA) membranes (Experimental)
  Interventions: Device: HDF with PMMA; Device: HDF
- patients on regular hemodialysis (HD) with polysulfone membrane dialyzers (HDF) (Active Comparator)
  Interventions: Device: HDF with PMMA; Device: HDF
- healthy individuals (No Intervention)

INTERVENTIONS:
Device: HDF with PMMA — Hemodiafiltration with polymethyl methacrylate (PMMA)-based membrane
  Arms: patients on regular hemodialysis (HD) HDF with high cut-off polymethylmethacrylate (PMMA) membranes; patients on regular hemodialysis (HD) with polysulfone membrane dialyzers (HDF)
Device: HDF — Hemodiafiltration without polymethyl methacrylate (PMMA)-based membrane
  Arms: patients on regular hemodialysis (HD) HDF with high cut-off polymethylmethacrylate (PMMA) membranes; patients on regular hemodialysis (HD) with polysulfone membrane dialyzers (HDF)

SUMMARY:
This is a randomized controlled crossover trial (58) in order to characterize PBL damage and death rate in hemodialysis patients treated with membranes with different permeability, including protein-leaking dialysers.

The study will enroll fourty patients on regular 4-h three times per week hemodialysis (HD) of the dialysis unit of the "Fondazione IRCCS Policlinico San Matteo" (Pavia, Italy). Thirteen age and sex matched healthy individuals (Ctr) and ten CKD patients on peritoneal dialysis treatment (PD*) will be included as healthy and CKD-matched controls, respectively. Comparison between HD and PD patients is aimed to assess the effect of biocompatibility and protein leakage during the treatments

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Male or female adults at time of enrolment aged <90 years old and >18 years old
* Patients in stable standard bicarbonate HD regimen, for at least two months

Exclusion Criteria:

* Patients aged <18 years old and >90 years old
* Known hypersensitivity or allergy to class of drugs or the investigational product or inability to comply with the requirements of the protocol;
* Participation in another study with investigational drug within the 30 days preceding and during the present study;
* Enrolment of the investigator, his/her family members, employees and other dependent persons;
* Recent illness (within the previous 1 week);
* Severe anemia (Hb < 7 g/dl);
* Bacterial or viral active infections;

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2027-02-17 (Estimated); Study Completion 2027-02-17 (Estimated)

PRIMARY OUTCOMES:
Comparison of the filters in term of the reduction of plasma HMWs and PBL death levels in a cross-over design | up to 24 months

SECONDARY OUTCOMES:
Identification of plasma proteins composition of the uremic retentates. | day 0, day 90, day 180
Pharmacological manipulation of the cellular redox in THP-1 human leukocytes exposed to uremic retention solutes. | day 0, day 90, day 180
  Thiol metabolomics and pharmacological manipulation of the cellular redox in THP-1 human leukocytes exposed to uremic retention solutes
Proteomics studies of the role of GSTP hyperexpression in the modulation of Nrf2 expression and activity in uremic leukocytes. | day 0, day 90, day 180
Study on transcription factors alternative to Nrf2 | day 0, day 90, day 180
  Study on transcription factors alternative to Nrf2 using human and murine Nrf2 inhibited monocyte lines
Study of Nrf2/GSTP stress response pathway in the PBL and THP-1 human monocytes | day 0, day 90, day 180
  Study of expression and activity of the Nrf2/GSTP stress response pathway in the PBL and THP-1 human monocytes exposed to isolated uremic retention solutes.
Study of cell death in PBL freshly isolated from study groups | day 0, day 90, day 180
  Study of cell death in PBL freshly isolated from study groups before and after treatment with autologous and heterologous whole plasma or isolated HMW fractions (studies of the IPR mechanism)
Analysis of CD4+ cells from blood samples and assessment of inflammatory cytokines after LPS stimulation | day 0, day 90, day 180
  Purification and culture of CD4+ cells from blood samples and assessment of inflammatory cytokines (IL-4, IL-10, IL-12 p70, IL-18, and IFNγ) after LPS stimulation
Determination of lymphocyte subpopulations ex vivo | day 0, day 90, day 180
Pathway analysis of the differentially expressed proteins of PBL and of principal component of complement system | day 0, day 90, day 180
Analysis of HMWs characteristic oxidative PTMs in plasma and PBL lysate samples collected | day 0, day 90, day 180

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia, Pavia, Italy